CLINICAL TRIAL: NCT03297515
Title: Prospective, Randomised, Double-blind Study to Assess the Therapeutic Potential of Omega-3 Fatty Acids Supplementation in Dry Macular Degeneration and Stargardt Disease (Macular Degeneration Omega-3 Study - MADEOS
Brief Title: Therapeutic Potential of Omega-3 Fatty Acids Supplementation in Dry Macular Degeneration and Stargardt Disease
Acronym: MADEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ophthalmos Research and Education Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG2017
Record Dates: First submitted 2017-09-22; First posted 2017-09-29 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Dry AMD; Stargardt Disease 1
Keywords: Omega-3; dry AMD; Stargardt; visual acuity
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega 3 fatty acids (Experimental): Omega 3 fatty acids
  Interventions: Dietary Supplement: Madeos
- Placebo (Placebo Comparator): Placebo (sunflower oil)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Madeos — Arm 1: Omega 3
  Arms: Omega 3 fatty acids
Dietary Supplement: Placebo — Arm 2 : Placebo
  Arms: Placebo

SUMMARY:
Prospective, randomised, double-blind study to assess the Therapeutic Potential of Omega-3 Fatty Acids Supplementation in Dry Macular Degeneration and Stargardt Disease (Macular Degeneration Omega-3 Study - MADEOS.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in developed countries. By the year 2040, the number of people suffering from AMD is estimated to increase by 50%. Stargardt disease is the most prevalent form of macular dystrophy in children, with an estimated prevalence of 1 in 10000.

There is no effective treatment available that stops progression or improves vision in patients with dry AMD or Stargardt disease.

Considering the success in animal studies and observational human studies with omega-3 fatty acids supplementation when the blood ratio AA (arachidonic acid)/EPA (eicosapentaenoic acid) is <2, the sponsor hypothesizes that, when the blood ratio of AA/EPA is maintained below 2, the visual acuity in the group with active supplements will improve, in comparison to the control group, in patients with moderate and severe dry AMD and moderate and severe Stargardt.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages from 18 to 85 years old.
* Group 1: For moderate dry macular degeneration the BCVA must be between 50 and 70 (ETDRS) at Screening Visit V1. There must be a large drusen >125 µm within 1mm from the centre of the fovea. Geographic atrophy can be present but must be >300 µm away from centre of fovea;
* Group 2: For severe dry macular degeneration the BCVA must be between 41 and 49 (ETDRS) at Screening Visit V1. Geographic atrophy can involve the fovea but must be <2500 µm in diameter or any size GA but >200 µm from centre of fovea anywhere;
* Group 3: For moderate Stargardt disease the BCVA must be between 50 and 70 (ETDRS) at Screening Visit V1. The geographic area must be <2.0 mm in diameter anywhere;
* Group 4: For severe Stargardt disease the BCVA must be between 41 and 49 (ETDRS) at Screening Visit V1. The geographic area must be <2.5 mm in diameter anywhere;
* Willingness to take the randomised trial investigational product for 6 months;
* Willingness to consent and undergo the examinations/blood testing at the visits;
* Be able to swallow large soft gel capsules;
* Take other supplements as usual; The EPA and DHA intake must be less than 1200 mg/day.

Exclusion Criteria:

* Any ocular disease in either eye including: Diabetic retinopathy, Central serous retinopathy, Epiretinal membrane, Optic atrophy, Macular hole or pseudohole, Retinal vein occlusion, Amblyopia;
* Previous wet AMD in the study eye;
* Any previous ocular surgery, which may influence progression of dry macular degeneration e.g. trabeculectomy, previous refractive surgery, pterygium surgery. Cataract surgery more than 6 months is not an exclusion criterion unless a complication has occurred during surgery;
* Any topical medication administered for other diseases such as glaucoma. Artificial tears up to 3/day will be allowed;
* Any ocular condition such as allergic conjunctivitis, moderate to severe dry eyes, scleritis, uveitis, keratitis, ocular Herpes Simplex keratitis, ectropion, entropion, ocular surface scaring;
* Any systemic conditions such as gastrointestinal disease e.g. irritable bowel syndrome, Crohn's disease, cancer, etc;
* Any drugs which could affect the eye administered up to 6 months before screening e.g.: Steroids, Ethambutol, Tamoxifen, Chloroquine, Hydroxychloroquine;
* Any condition that would not allow follow up e.g. alcoholism or drug abuse;
* Allergy to any ingredients of the active or placebo pills.
* Pregnant or lactating;
* Current use of EPA/DHA supplements in excess of 1200 mg/day;
* History of liver disease;
* Anti-coagulation therapy such as warfarin/heparin/aspirin/dabigatran/ clopidogrel etc;
* Bleeding tendencies e.g. coagulopathies;
* History of atrial fibrillation;
* Inability to give informed consent (impaired mental capacity e.g. psychiatric deficit);
* Smokers or patients who have not been completely smoke free over the past 5 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Mean change of letters (BCVA) from screening to 24 weeks | 24 weeks
  Mean change of letters (BCVA) from screening to 24 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Centre National d'Ophtalmologie des Quinze-Vingts, Paris, France
- Department of Ophthalmology, Justus-Liebig-University-Giessen, Giessen, Germany
- Italy (3):
  - Università degli Studi G. d'Annunzio Chieti-Pescara, Chieti
  - ASST Santi Paolo e Carlo, Milan
  - Department of Ophthalmology, University Vita Salute, Milan